CLINICAL TRIAL: NCT04798742
Title: Gluteus Maximus Transfer Following THA Does Not Improve Abductor Strength - a Case-control Gait Analysis Study of 15 Patients With Gluteus Medius Disruption
Brief Title: Gluteus Maximus Transfer Following THA Does Not Improve Abductor Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Gluteus maximus transfer
Record Dates: First submitted 2021-02-24; First posted 2021-03-15 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait performance preop vs postop (Experimental): Pre and postop
  Interventions: Procedure: Gluteus maximus transfer
- Gait performance postop vs controls (Experimental): Postop vs controls
  Interventions: Procedure: Gluteus maximus transfer

INTERVENTIONS:
Procedure: Gluteus maximus transfer — Gait analysis study of 15 patients with gluteus medius disruption

SUMMARY:
Gluteus maximus transfer following THA does not improve abductor strength - a case-control gait analysis study of 15 patients with gluteus medius disruption

The investigators have compared 15 gluteus maximus transferred patients with the use of a gait analysis system based on reflective markers and force plates to objectively evaluate the gait performance pre- and postoperatively.

DETAILED DESCRIPTION:
The gluteus maximus flap transfer (GMT) is a surgical technique to improve gait kinematics and kinetics as well as reduce pain and ameliorate functional outcome in patients with hip abductor deficiency of the gluteus medius following total hip arthroplasty (THA). The investigators used a gait analysis system based on reflective markers and force plates to objectively evaluate gait performance pre- and postoperatively.

Methods Gait analysis was performed in 15 patients who underwent GMT and were examined with an optical tracking system before and at a minimum of 13 months after the operation. Mean age was 69 years (SD=11), all were females. Median follow-up time was 24 (13-60) months. The primary outcome was hip abduction moment (Nm/kg) during gait. The control group consisted of 66 subjects without any gait pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip abductor deficiency of the gluteus medius following total hip arthroplasty (THA)

Exclusion Criteria:

* THA prior to the muscle transfer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Abductor strength measurement with use of an optical tracking system after Gluteus maximus transfer - a case-control gait analysis study of 15 patients pre- and postoperative with gluteus medius disruption | Preop
  Gait analysis examination/measure will be performed preoperative with an optical tracking system in a gait laboratory using reflective markers and integrated force plates in order to record kinetics (Nm/kg) of abductor muscles moment in the frontal plane.
Abductor strength measurement with use of an optical tracking system after Gluteus maximus transfer- a case-control gait analysis study of 15 patients pre- and postoperative with gluteus medius disruption | Postop 2 year
  Gait analysis examination/measure will be performed 2 year postoperative with an optical tracking system in a gait laboratory using reflective markers and integrated force plates in order to record kinetics (Nm/kg) of abductor muscles moment in the frontal plane.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zügner, Principal Investigator — Göteborg University
Locations (1):
- Roland Zügner, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After publication, all available data will be available by appointment and within a reasonable time.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication and 2 years after publication

REFERENCES:
- [Result] Whiteside LA. Surgical technique: Transfer of the anterior portion of the gluteus maximus muscle for abductor deficiency of the hip. Clin Orthop Relat Res. 2012 Feb;470(2):503-10. doi: 10.1007/s11999-011-1975-y. PMID 21796476